CLINICAL TRIAL: NCT00346086
Title: A Phase II Observer-blind, Randomized, Placebo-Controlled Study of the Efficacy, Safety, Tolerability, and Immunogenicity of Subcutaneously Administered Dynavax Amb a 1 Immunostimulatory Oligodeoxyribonucleotide Conjugate (AIC) in Ragweed-Allergic Adults (Sponsor's Protocol NRH01)
Brief Title: DNA Vaccine for Ragweed Allergic Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAC01-03-27-01; NRH01
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: CpG oligonucleotide vaccine; ragweed immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Aminoimidazole Carboxamide

INTERVENTIONS:
Drug: AIC (Amb a 1 Immunostimulatory Conjugate)

SUMMARY:
Various chemical modifications of allergens have been attempted to enhance efficacy, improve safety, and foster compliance with IT. These approaches have been unsuccessful - in that the allergenicity and immunogenicity have either decreased, or increased in tandem, with no resultant efficacy: safety benefit ratio. This study utilizes an adjuvant approach in which synthetic immunostimulatory DNA is conjugated to ragweed allergen in an attempt to modulate both the clinical and immunologic allergic response to ragweed exposure in ragweed-allergic patients with seasonal rhinitis.

DETAILED DESCRIPTION:
Evaluation of efficacy and safety of allergen-CpG oligonucleotide immunostimulatory conjugate in treatment of ragweed-induced seasonal allergic rhinitis. Study incorporates clinical outcomes (symptom diaries, medication diaries, visual analog scores, quality of life questionnaires), safety measurements, immunologic assays (antibody measurements, T-cell assays, cytokine assays, nasal provocation).

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women 18 to 60 years of age;
* Who provide informed consent;
* Have a history of fall, seasonal, allergic rhinitis consistent with ragweed allergy;
* Exhibit a positive skin test to licensed , standardized, ragweed extract and a positive acute response to ragweed nasal challenge;
* Are in general good health; and are available for the duration of the study.

Exclusion Criteria:

* Individuals with medical conditions or taking medications that might interfere with interpretation of the study results will be excluded.
* Those with a history of severe symptoms of allergic rhinitis during the spring and summer grass pollen season will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2001-05-18 (Actual); Primary Completion 2001-08-21 (Actual); Study Completion 2001-08-21 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on nasal allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Creticos, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Creticos PS, Schroeder JT, Hamilton RG, Balcer-Whaley SL, Khattignavong AP, Lindblad R, Li H, Coffman R, Seyfert V, Eiden JJ, Broide D; Immune Tolerance Network Group. Immunotherapy with a ragweed-toll-like receptor 9 agonist vaccine for allergic rhinitis. N Engl J Med. 2006 Oct 5;355(14):1445-55. doi: 10.1056/NEJMoa052916. PMID 17021320